CLINICAL TRIAL: NCT04109040
Title: Patients' Satisfaction After LASIK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Sayed Mohamed, post gradute doctor, Assiut University
Other Study IDs: LASIK
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Slit Lamp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: slit lamp — diagnostice device to examine anterior segment of the eye and for fundus examination

SUMMARY:
The aim of this study is to evaluate the level of satisfaction, functional vision and quality of life outcome of patients after LASIK surgery.

DETAILED DESCRIPTION:
The feeling of sight in human is usually taken as the most significant factor for fathoming and receiving data from environment and, thus, assumes a significant role in regulating most human exercises and practices. Accordingly, any harm to this sense may significantly influence an individual's adjustment with environment.1

Refractive error can be explained as an eye condition in which incoming light rays are not focused on the photoreceptor layer of the fovea, resulting in blurred vision. Of the refractive errors, myopia, hyperopia, and astigmatism are the 3 most common types. In myopia, the incoming light rays are focused in front of the fovea, whereas in hyperopia, they are focused beyond the fovea. Astigmatism is typically explained by irregularities in the cornea (corneal astigmatism) and crystalline lens (lenticular astigmatism), which results in differential focusing of parallel rays through different corneal and lenticular meridians.The refractive surgery has a very important role helping subjects to get rid of contact lenses and spectacules.2-3

Laser-assisted in situ keratomileusis (LASIK) is the most popular refractive surgery performed to correct refractive errors of the eye, including myopia, hyperopia, and astigmatism. LASIK surgery has been reported to yield significantly improved patient reported visual outcomes.1 The result is the patient's independence from glasses and contact lenses. Many studies have reported that LASIK surgery can improve not only visual function,1 but also patients' quality of life (QOL).2,4-10

Patient-reported outcomes also revealed that LASIK can maximize patient satisfaction and quality of life by minimizing the onset of visual and dry eye symptoms.11 Happiness or positive emotions are now regarded as a critical component of health.12 With the introduction of the discipline of positive psychology in the late 1990s, many scientific investigations of happiness have resulted in the development of the proposal that happiness or positive emotions are highly beneficial for physical and mental health.12-19

ELIGIBILITY:
Inclusion Criteria:

Patients with myopia less than -10 Diopters Patients with hyperopia less than + 6 Diopters

Exclusion Criteria:

Patients of eye disease that may interfere with the results of the study. Previous ocular surgery. Patients using psychiatric medication will not be included in the study. Unwillingness to participate in the study. Subjects who did not respond to all questions were excluded.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The study population included were both males and females in private LASIK center . The inclusion criteria are patients who have suffered from refractive errors aged from 18 - 55years old and patients who have done LASIK within one year for at least 3 monthes will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
patients' satisfaction after LASIK | LASIK
  to evaluate the level of satisfaction and quality of life outcome of patients after LASIK surgery and funtional vision to improve quality of life and help patients to get rid of glasses

REFERENCES:
- [Background] Hays RD, Tarver ME, Spritzer KL, Reise S, Hilmantel G, Hofmeister EM, Hammel K, May J, Ferris F 3rd, Eydelman M. Assessment of the Psychometric Properties of a Questionnaire Assessing Patient-Reported Outcomes With Laser In Situ Keratomileusis (PROWL). JAMA Ophthalmol. 2017 Jan 1;135(1):3-12. doi: 10.1001/jamaophthalmol.2016.4597. PMID 27893063